CLINICAL TRIAL: NCT02423993
Title: Efficiency Assessment of the Structured Education Program for Type 1 Diabetes Patients on Insulin Pump Therapy
Brief Title: Education Effectiveness for Type 1 Diabetes Mellitus on Insulin Pump Therapy
Acronym: EASEDIAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Endocrinology Research Centre, Moscow (Other Government)
Responsible Party: Principal Investigator, Ibragimova Lyudmila, MD, PhD, Endocrinology Research Centre, Moscow
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 101-01-2010
Record Dates: First submitted 2015-04-19; First posted 2015-04-22 (Estimated); Results first posted 2016-01-11 (Estimated); Last update posted 2016-01-11 (Estimated); Status verified 2015-12

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: Type 1 diabetes mellitus; Continuous subcutaneous insulin infusion; Quality of life; Therapeutic education; Insulin pump
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Mass Screening

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- SAP + Group Education (Experimental): Patients will be transferred from MDI to sensor-augmented pump (SAP) in group using specialised structured education program. CGM will be used for self monitoring of blood glucose permanently within 4 month.
  Interventions: Behavioral: Education by structured programme; Device: CSII; Device: CGM-RT; Procedure: Screening for Complications; Procedure: Glycaemic control assessment; Procedure: QoL assessment; Procedure: Knowledge assessment
- SAP + Standard Education (Active Comparator): Patients will be transferred from MDI to sensor-augmented pump (SAP) by endocrinologist-specialist in CSII or technical trainer individually and will be monitored by coaching specialist or local endocrinologist within 4 months prior to inclusion. All patients from this group should be educated about basic aspects of diabetes self-management at the School of Diabetes at least once earlier.
  Interventions: Device: CSII; Device: CGM-RT; Procedure: Screening for Complications; Procedure: Glycaemic control assessment; Procedure: QoL assessment; Procedure: Knowledge assessment
- CSII + Group Education (Experimental): Patients will be transferred from MDI to CSII with self-monitoring of blood glucose (SMBG) using specialised structured education program.
  Interventions: Behavioral: Education by structured programme; Device: CSII; Procedure: Screening for Complications; Procedure: Glycaemic control assessment; Procedure: QoL assessment; Procedure: Knowledge assessment
- CSII + Standard Education (Active Comparator): Patients will be transferred from MDI to CSII with self-monitoring of blood glucose (SMBG) by endocrinologist-specialist in CSII or technical trainer individually and will be monitored by coaching specialist or local endocrinologist within 4 months prior to inclusion. All patients from this group should be educated about basic aspects of diabetes self-management at the School of Diabetes at least once earlier.
  Interventions: Device: CSII; Procedure: Screening for Complications; Procedure: Glycaemic control assessment; Procedure: QoL assessment; Procedure: Knowledge assessment

INTERVENTIONS:
Behavioral: Education by structured programme — Thе structured programme was developed in Endocrinology Research Centre. It is based on the following principles: education in group setting, using structured program; intensive insulin treatment using insulin pumps; self-adjustment of insulin dose and pump settings; intensive self-monitoring of blood glucose, including continuous glucose monitoring in real-time ("CGM-RT"); flexible physical activities and meals regimen (liberal diet, based on carbohydrates account using bread units; possible shifts of meals schedule and volume supported by appropriate treatment adjustment). Duration of education course - 8 days (35-37 hours); planned group volume is 7-10 patients.
  Arms: CSII + Group Education; SAP + Group Education
Device: CSII — The intensified insulin therapy by means of continuous subcutaneous insulin infusion will be provide by Medtronic insulin pumps: Paradigm MMT-712/715, Paradigm Real-Time MMT-722, Paradigm VEO MMT-754.
Device: CGM-RT — Continuous glucose monitoring ("CGM") will be provide by means of Paradigm Real-Time MMT-722 and Paradigm VEO MMT-754 Medtronic sensor-augmented insulin pumps. For monitoring the Sof-Sensor and MiniLink transmitter (Medtronic) will be use. Each sensor will be use for 6 days. CGM will be use for self-monitoring of blood glucose on permanent basis (more than 6 days per week) within 4 month.
  Arms: SAP + Group Education; SAP + Standard Education
Procedure: Screening for Complications — To assess diabetic retinopathy a fundoscopy will be held. Diabetic nephropathy will be assessed by microalbuminuria screening, serum creatinine evaluation and calculation of CKD-EPI glomerular filtration rate. Diabetic neuropathy will be assessed by all kinds of sensitivity evaluation (vibrating, tactile, temperature).
Procedure: Glycaemic control assessment — Glycemic control effectiveness changes will be assessed by measure of glycated hemoglobin (HbA1c). The frequency of blood glucose self-monitoring will be estimated by patient's diaries evaluation, individual glucometer data evaluation and insulin pump reports. Bolus calculator use and hypoglycemia nonsevere frequency will be assessed by reports received from insulin pumps.
Procedure: QoL assessment — For Quality of Life ("QoL") assessment will be used the following validated questionnaires (in Russian):
  1. The Medical Outcomes Study 36-Item Short Form Health Survey - SF-36.
  2. The Audit of the Diabetes-Dependent Quality of Life - ADDQoL (С. Bradley et al, 1999, adjusted by Starostina E.G., 2003).
Procedure: Knowledge assessment — For the knowledge assessment of disease management the standard Questionnaire for patients with type 1 diabetes will be used. Maximum score equals 37 grades; the satisfactory level of knowledge is scored 27.

SUMMARY:
The purpose of this study is to assess the effectiveness of structured group education on glycemic control and Quality of Life (QoL) among users of continuous subcutaneous insulin infusions (CSII).

DETAILED DESCRIPTION:
The study will include 80 patients with type 1 diabetes that will be transferred from multiple daily injection (MDI) regimen to continuous subcutaneous insulin infusion (CSII). All patients will be divided into 2 groups: 1) structured education group (n=40) and 2) control group (n=40).

Patients from structured education group will be transferred from MDI to CSII using special structured education program for type 1 diabetes patients on insulin pump therapy. Before the transferring to CSII the patients from this group will be randomized in two subgroups, depending on type of blood glucose control: patients which will use CSII and self-monitoring of blood glucose (SMBG) (n=20) or patients which will use sensor-augmented pump (SAP) (n=20).

Follow-up duration in structured education group will be 4 months; follow-up visits included treatment adjustment, glucose data review and and collection of data on adverse events every 4 weeks. Between visits, communication with clinicians will be initiated at the discretion of the patient.

The control group will include patients with type 1 diabetes using CSII during 4-6 months before. The patients from this group will be divided in two subgroups, depending on type of self blood glucose control: patients using CSII (n=20) and SMBG or patients using SAP (n=20). In this group patients should be transferred to CSII by endocrinologist-specialist in CSII or technical trainer individually and will be monitored by coaching specialist or local endocrinologist within 4 months prior to inclusion. All patients from this group should be educated in intensive diabetes management, including carbohydrate counting, the administration of correction doses of insulin and technical aspects of CSII and self glucose control by continuous glucose monitoring in real-time ("CGM-RT").

All patients will provide written informed consent.

Diabetes-management software (CareLink Therapy Management System for Diabetes-Clinical, Medtronic) will be used for glucose data review including frequency of hypoglycemia, assessment of frequency of bolus calculator use.

Diaries of self-control will be analysed for glucose data review.

The level of knowledge about the basics of diabetes self-management will be assessed using a standard questionnaire for patients with type 1 diabetes.

For Quality of Life (QoL) assessment will be used the following validated questionnaires (in Russian):

1. The Medical Outcomes Study 36-Item Short Form Health Survey (SF-36).
2. The Audit of the Diabetes-Dependent Quality of Life (ADDQoL) (С. Bradley et al., 1999, adjusted by Starostina E.G., 2003).

Patients from structured education group will complete the QoL Questionnaires prior to education and 4 months after transferring to CSII. Patients from the control group will complete the Questionnaires during the enrollment.

Assessment of diabetes complications will be held before and 4 months after transferring to CSII in structured education group and at the time of enrollment in control group.

For the knowledge assessment of disease management will be used standard Questionnaire for patients with type 1 diabetes. Maximum score equals 37 grades; the satisfactory level of knowledge is scored 27. Patients from the structural education group will complete the Questionnaire prior to conversion to CSII regimen and the education course and after 4 months of the follow up. Patients from the control group will complete the Questionnaire during enrollment.

Statistical analysis. Statistica (StatSoft Inc., USA, version 8.0) software will be used for data processing. The following descriptive statistical parameters will be used: median, inter-quartile interval (Me [25;75]) and mass share (%). Non- parametric criteria will be used used for non-normalized distribution (Mann - Whitney U-criterion for paired comparison of independent samples). The χ2 criterion was used for comparison of parameters distribution in population samples. Non - parametric Spearman's correlation will be used for correlation analysis. Standard deviation (M±SD) will be used to evaluate the rate of hypoglycemia events, frequency of plasma glucose level self-control, utilization of bolus calculator, plasma glucose level variability, and for certain items of QoL Questionnaires. A P value of less than 0.05 will be considered to indicate statistical significance for comparisons of the primary outcome, baseline characteristics, and safety.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes mellitus;
* Disease duration > 1 year;
* Patients informed consent, approving participation and completion of questionnaires.

Exclusion Criteria:

* Severe late diabetic complications (diabetic foot syndrome, painful neuropathy, autonomic neuropathy, significant loss of vision, glomerular filtration rate < 30 ml/min/1.73 m2);
* Pregnancy;
* Severe concomitant diseases;
* Known psychic disorders and/or treatment with psychotropic medicines.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2009-10; Primary Completion 2012-10 (Actual); Study Completion 2013-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aleksandr Y Mayorov, MD,PhD, Study Chair — Endocrinology Research Centre; Marina V Shestakova, MD,PhD,Prof, Study Director — Endocrinology Research Centre; Lyudmila I Ibragimova, MD, PhD, Principal Investigator — Endocrinology Research Centre

REFERENCES:
- [Background] Effect of intensive diabetes treatment on the development and progression of long-term complications in adolescents with insulin-dependent diabetes mellitus: Diabetes Control and Complications Trial. Diabetes Control and Complications Trial Research Group. J Pediatr. 1994 Aug;125(2):177-88. doi: 10.1016/s0022-3476(94)70190-3. PMID 8040759
- [Background] Bradley C, Speight J. Patient perceptions of diabetes and diabetes therapy: assessing quality of life. Diabetes Metab Res Rev. 2002 Sep-Oct;18 Suppl 3:S64-9. doi: 10.1002/dmrr.279. PMID 12324988
- [Background] Clark M. Diabetes self-management education: a review of published studies. Prim Care Diabetes. 2008 Sep;2(3):113-20. doi: 10.1016/j.pcd.2008.04.004. Epub 2008 Jun 25. PMID 18779034
- [Background] Corriveau EA, Durso PJ, Kaufman ED, Skipper BJ, Laskaratos LA, Heintzman KB. Effect of Carelink, an internet-based insulin pump monitoring system, on glycemic control in rural and urban children with type 1 diabetes mellitus. Pediatr Diabetes. 2008 Aug;9(4 Pt 2):360-6. doi: 10.1111/j.1399-5448.2008.00363.x. PMID 18774996
- [Background] Gross TM, Kayne D, King A, Rother C, Juth S. A bolus calculator is an effective means of controlling postprandial glycemia in patients on insulin pump therapy. Diabetes Technol Ther. 2003;5(3):365-9. doi: 10.1089/152091503765691848. PMID 12828818
- [Background] DAFNE Study Group. Training in flexible, intensive insulin management to enable dietary freedom in people with type 1 diabetes: dose adjustment for normal eating (DAFNE) randomised controlled trial. BMJ. 2002 Oct 5;325(7367):746. doi: 10.1136/bmj.325.7367.746. PMID 12364302
- [Background] Home PD, Pickup JC, Keen H, Alberti KG, Parsons JA, Binder C. Continuous subcutaneous insulin infusion: comparison of plasma insulin profiles after infusion or bolus injection of the mealtime dose. Metabolism. 1981 May;30(5):439-42. doi: 10.1016/0026-0495(81)90177-3. PMID 6112654
- [Background] Lauritzen T, Pramming S, Deckert T, Binder C. Pharmacokinetics of continuous subcutaneous insulin infusion. Diabetologia. 1983 May;24(5):326-9. doi: 10.1007/BF00251817. PMID 6347780
- [Background] Ludwig-Seibold CU, Holder M, Rami B, Raile K, Heidtmann B, Holl RW; DPV Science Initiative; German Working Group for insulin pump treatment in pediatric patients; German BMBF Competence Network Diabetes. Continuous glucose monitoring in children, adolescents, and adults with type 1 diabetes mellitus: analysis from the prospective DPV diabetes documentation and quality management system from Germany and Austria. Pediatr Diabetes. 2012 Feb;13(1):12-4. doi: 10.1111/j.1399-5448.2011.00835.x. Epub 2011 Nov 29. PMID 22128781
- [Background] Misso ML, Egberts KJ, Page M, O'Connor D, Shaw J. Continuous subcutaneous insulin infusion (CSII) versus multiple insulin injections for type 1 diabetes mellitus. Cochrane Database Syst Rev. 2010 Jan 20;2010(1):CD005103. doi: 10.1002/14651858.CD005103.pub2. PMID 20091571
- [Background] Nixon R, Pickup JC. Fear of hypoglycemia in type 1 diabetes managed by continuous subcutaneous insulin infusion: is it associated with poor glycemic control? Diabetes Technol Ther. 2011 Feb;13(2):93-8. doi: 10.1089/dia.2010.0192. PMID 21284474
- [Background] Pedersen-Bjergaard U, Pramming S, Heller SR, Wallace TM, Rasmussen AK, Jorgensen HV, Matthews DR, Hougaard P, Thorsteinsson B. Severe hypoglycaemia in 1076 adult patients with type 1 diabetes: influence of risk markers and selection. Diabetes Metab Res Rev. 2004 Nov-Dec;20(6):479-86. doi: 10.1002/dmrr.482. PMID 15386817
- [Background] Pickup JC, Keen H, Parsons JA, Alberti KG. Continuous subcutaneous insulin infusion: an approach to achieving normoglycaemia. Br Med J. 1978 Jan 28;1(6107):204-7. doi: 10.1136/bmj.1.6107.204. PMID 340000
- [Background] Rubin RR, Borgman SK, Sulik BT. Crossing the technology divide: practical strategies for transitioning patients from multiple daily insulin injections to sensor-augmented pump therapy. Diabetes Educ. 2011 Jan-Feb;37 Suppl 1:5S-18S; quiz 19S-20S. doi: 10.1177/0145721710391107. Epub 2011 Jan 7. PMID 21217102
- [Background] Rubin RR, Peyrot M. Quality of life and diabetes. Diabetes Metab Res Rev. 1999 May-Jun;15(3):205-18. doi: 10.1002/(sici)1520-7560(199905/06)15:33.0.co;2-o. PMID 10441043
- [Background] Riveline JP. Is continuous glucose monitoring (CGM) for everyone? To whom should CGM be prescribed and how? Diabetes Metab. 2011 Dec;37 Suppl 4:S80-4. doi: 10.1016/S1262-3636(11)70971-5. PMID 22208716
- [Background] Schwartz FL, Guo A, Marling CR, Shubrook JH. Analysis of use of an automated bolus calculator reduces fear of hypoglycemia and improves confidence in dosage accuracy in type 1 diabetes mellitus patients treated with multiple daily insulin injections. J Diabetes Sci Technol. 2012 Jan 1;6(1):150-2. doi: 10.1177/193229681200600118. PMID 22401333
- [Background] Shashaj B, Busetto E, Sulli N. Benefits of a bolus calculator in pre- and postprandial glycaemic control and meal flexibility of paediatric patients using continuous subcutaneous insulin infusion (CSII). Diabet Med. 2008 Sep;25(9):1036-42. doi: 10.1111/j.1464-5491.2008.02549.x. PMID 18937673
- [Background] Wu YP, Graves MM, Roberts MC, Mitchell AC. Is insulin pump therapy better than injection for adolescents with diabetes? Diabetes Res Clin Pract. 2010 Aug;89(2):121-5. doi: 10.1016/j.diabres.2010.04.010. Epub 2010 May 21. PMID 20488572
- [Background] Philippov YI. Continuous monitoring of blood glucose in the practice of endocrinologist. Obesity and metabolism 9(4):15-22, 2012. doi: 10.14341/2071-8713-5124
- [Background] Filippov YI, Pekareva EV, Mayorov AY. Selected aspects of insulin pump therapy and continuous glucose monitoring in real time ( in relation to the letter of E.D.Gorbachev). Diabetes mellitus 13(4):119-124, 2010. doi: 10.14341/2072-0351-6074
- [Result] Ibragimova LI, Filippov YI, Mayorov AY. Insulin pump therapy in type 1 diabetes mellitus: education effectiveness and quality of life. Diabetes mellitus 15(1):35-40, 2012. doi: 10.14341/2072-0351-5977
- See also: Endocrinology Research Centre — http://www.endocrincentr.ru/

RESULTS

PARTICIPANT FLOW:
Groups:
- SAP + Group Education: All patients were transferred from MDI regimen to sensor-augmented pump (Medtronic Paradigm Real-Time MMT-722, Paradigm VEO MMT-754.) using special structured program for group education for CSII which included basic information about general diabetes self-management and technical aspects of pump therapy for 9 days. QoL was assessed using questionnaire ADDQoL, WB12, SF-36. Glycemic control effectiveness changes were assessed by measure of glycated hemoglobin (HbA1c). The frequency of blood glucose self-monitoring was estimated by patient's diaries evaluation, individual glucometer data evaluation and insulin pump reports. Bolus calculator use and hypoglycemia nonsevere frequency was assessed by reports received from insulin pumps. Standard Questionnaire for patients with type 1 diabetes was used for the knowledge assessment about disease management.
  We estimated metabolic and QoL parameters in 4 months after education and transferring to CSII.
- SAP + Standart Education: Patients were transferred from MDI to sensor-augmented pump (Medtronic Paradigm Real-Time MMT-722) by endocrinologist-specialist in CSII or technical trainer individually and will be monitored by coaching specialist or local endocrinologist within 4 months prior to inclusion. CGM was used for self-monitoring of blood glucose on permanent basis (more than 6 days per week) within 4 months. All patients from this group were educated about basic aspects of diabetes self-management earlier. QoL was assessed using questionnaire ADDQoL, WB12, SF-36. Glycemic control effectiveness changes was assessed by HbA1c. The frequency of blood glucose self-monitoring was estimated by patient's diaries evaluation, individual glucometer data evaluation and insulin pump reports. Bolus calculator use and hypoglycemia nonsevere frequency were assessed by reports received from insulin pumps. Standard Questionnaire for patients with T1D was used for the knowledge assessment about disease management.
- CSII + Group Education: Patients was transferred from MDI to CSII (Medtronic Paradigm 712) with self-monitoring of blood glucose (SMBG) using specialised structured education program for group education for CSII which included basic information about general diabetes self-management and technical aspects of pump therapy for 9 days. Quality of Life was assessed using questionnaire ADDQoL, WB12, SF-36. Glycemic control effectiveness changes was assessed by measure of glycated hemoglobin (HbA1c). The frequency of blood glucose self-monitoring was estimated by patient's diaries evaluation, individual glucometer data evaluation and insulin pump reports. Bolus calculator use and hypoglycemia nonsevere frequency were assessed by reports received from insulin pumps. Knowledge assessment of disease management the standard Questionnaire for patients with type 1 diabetes was used.
  We estimated metabolic and QoL parameters in 4 months after education and transferring to CSII.
- CSII + Standart Education: Patients were transferred from MDI to CSII (Medtronic Paradigm 712) with self-monitoring of blood glucose (SMBG) by endocrinologist-specialist in CSII or technical trainer individually and were monitored by coaching specialist or local endocrinologist within 4 months prior to inclusion. All patients from this group were educated about basic aspects of diabetes self-management earlier. Quality of Life (QoL) was assessed using questionnaire ADDQoL, WB12, SF-36. Glycemic control effectiveness changes were assessed by measure of glycated hemoglobin (HbA1c). The frequency of blood glucose self-monitoring was estimated by patient's diaries evaluation, individual glucometer data evaluation and insulin pump reports. Bolus calculator use and hypoglycemia nonsevere frequency were assessed by reports received from insulin pumps. Knowledge assessment of disease management the standard Questionnaire for patients with type 1 diabetes was used.
Period: Overall Study
Arm/Group | SAP + Group Education | SAP + Standart Education | CSII + Group Education | CSII + Standart Education
Started | 19 | 16 | 23 | 19
Completed | 19 | 16 | 23 | 19
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- SAP + Group Education: All patients will be transferred from MDI regimen to sensor-augmented pump (Medtronic Paradigm Real-Time MMT-722, Paradigm VEO MMT-754) using special structured program for group education for CSII which included basic information about general diabetes self-management and technical aspects of pump therapy for 9 days. Quality of Life will be assessed using questionnaire ADDQoL, WB12, SF-36. Glycemic control effectiveness changes will be assessed by measure of glycated hemoglobin (HbA1c). The frequency of blood glucose self-monitoring will be estimated by patient's diaries evaluation, individual glucometer data evaluation and insulin pump reports. Bolus calculator use and hypoglycemia nonsevere frequency will be assessed by reports received from insulin pumps. Knowledge assessment of disease management the standard Questionnaire for patients with type 1 diabetes will be used.
  We will estimate metabolic and QoL parameters in 4 months after education and transferring to CSII.
- SAP + Standart Education: Patients will be transferred from MDI to sensor-augmented pump (Medtronic Paradigm Real-Time MMT-722, Paradigm VEO MMT-754) by endocrinologist-specialist in CSII or technical trainer individually and will be monitored by coaching specialist or local endocrinologist within 4 months prior to inclusion. CGM will be used for self-monitoring of blood glucose on permanent basis (more than 6 days per week) within 4 month. All patients from this group should be educated about basic aspects of diabetes self-management at the School of Diabetes at least once earlier. Quality of Life (QoL) will be assessed using questionnaire ADDQoL, WB12, SF-36. Glycemic control effectiveness changes will be assessed by measure of glycated hemoglobin (HbA1c). The frequency of blood glucose self-monitoring will be estimated by patient's diaries evaluation, individual glucometer data evaluation and insulin pump reports. Bolus calculator use and hypoglycemia nonsevere frequency will be assessed by reports received
- CSII + Group Education: Patients will be transferred from MDI to CSII with self-monitoring of blood glucose (SMBG) using specialised structured education program for group education for CSII which included basic information about general diabetes self-management and technical aspects of pump therapy for 9 days. Quality of Life will be assessed using questionnaire ADDQoL, WB12, SF-36. Glycemic control effectiveness changes will be assessed by measure of glycated hemoglobin (HbA1c). The frequency of blood glucose self-monitoring will be estimated by patient's diaries evaluation, individual glucometer data evaluation and insulin pump reports. Bolus calculator use and hypoglycemia nonsevere frequency will be assessed by reports received from insulin pumps. Knowledge assessment of disease management the standard Questionnaire for patients with type 1 diabetes will be used.
  We will estimate metabolic and QoL parameters in 4 months after education and transferring to CSII.
- CSII + Standart Education: Patients will be transferred from MDI to CSII (Medtronic Paradigm 712) with self-monitoring of blood glucose (SMBG) by endocrinologist-specialist in CSII or technical trainer individually and will be monitored by coaching specialist or local endocrinologist within 4 months prior to inclusion. All patients from this group should be educated about basic aspects of diabetes self-management at the School of Diabetes at least once earlier. Quality of Life (QoL) will be assessed using questionnaire ADDQoL, WB12, SF-36. Glycemic control effectiveness changes will be assessed by HbA1c. The frequency of blood glucose self-monitoring will be estimated by patient's diaries evaluation, individual glucometer data evaluation and insulin pump reports. Bolus calculator use and hypoglycemia nonsevere frequency will be assessed by reports received from insulin pumps. Knowledge assessment of disease management the standard Questionnaire for patients with type 1 diabetes will be used.
- Total: Total of all reporting groups
Arm/Group | SAP + Group Education | SAP + Standart Education | CSII + Group Education | CSII + Standart Education | Total
Number analyzed (Participants) | 19 | 16 | 23 | 19 | 77
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 19 | 16 | 23 | 19 | 77
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 29.5 [29 to 36] | 33 [25 to 36] | 27 [25 to 35] | 23 [19 to 28] | 26.5 [24 to 36]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 8 | 14 | 11 | 44
  Male | 8 | 8 | 9 | 8 | 33
Region of Enrollment [Number; unit: participants]
  Russian Federation | 19 | 16 | 23 | 19 | 77

OUTCOME MEASURES:

1. Primary Outcome: HbA1c
Description: HbA1c was determined by ion exchange chromatography on an automatic biochemical analyzer Bio-RAD D-10 (France), under the manufacturer's standard procedure.
Time Frame: 4 month after CSII initiation
Population: The analysis was "per protocol". Patients from group education groups were on MDI regymen and from standart education group were on insulin pump therapy during previously 4 months
Measure: Median (Inter-Quartile Range); unit: percentage
Groups:
- SAP + Standard Education: Patients were transferred from MDI to sensor-augmented pump (Medtronic Paradigm Real-Time MMT-722) by endocrinologist-specialist in CSII or technical trainer individually and will be monitored by coaching specialist or local endocrinologist within 4 months prior to inclusion. CGM was used for self-monitoring of blood glucose on permanent basis (more than 6 days per week) within 4 months. All patients from this group were educated about basic aspects of diabetes self-management earlier. QoL was assessed using questionnaire ADDQoL, WB12, SF-36. Glycemic control effectiveness changes was assessed by HbA1c. The frequency of blood glucose self-monitoring was estimated by patient's diaries evaluation, individual glucometer data evaluation and insulin pump reports. Bolus calculator use and hypoglycemia nonsevere frequency were assessed by reports received from insulin pumps. Standard Questionnaire for patients with T1D was used for the knowledge assessment about disease management.
- CSII + Standard Education: Patients were transferred from MDI to CSII (Medtronic Paradigm 712) with self-monitoring of blood glucose (SMBG) by endocrinologist-specialist in CSII or technical trainer individually and were monitored by coaching specialist or local endocrinologist within 4 months prior to inclusion. All patients from this group were educated about basic aspects of diabetes self-management earlier. Quality of Life (QoL) was assessed using questionnaire ADDQoL, WB12, SF-36. Glycemic control effectiveness changes were assessed by measure of glycated hemoglobin (HbA1c). The frequency of blood glucose self-monitoring was estimated by patient's diaries evaluation, individual glucometer data evaluation and insulin pump reports. Bolus calculator use and hypoglycemia nonsevere frequency were assessed by reports received from insulin pumps. Knowledge assessment of disease management the standard Questionnaire for patients with type 1 diabetes was used.
Arm/Group | SAP + Group Education | SAP + Standard Education | CSII + Group Education | CSII + Standard Education
Number analyzed (Participants) | 19 | 16 | 23 | 19
percentage | 7.3 [6.3 to 7.8] | 8.0 [6.3 to 8.5] | 7.5 [6.9 to 8.2] | 8.8 [8.0 to 9.7]

2. Secondary Outcome: Severe Hypoglycaemia Frequency
Description: Severe hypoglycemia is defined аs an episode requiring assistance and will be confirmed by documentation of a blood glucose value of less than 50 mg per deciliter (2.8 mmol per liter) or recovery with restoration of plasma glucose.
Time Frame: within 4 month of the study
Measure: Mean (Standard Deviation); unit: events per month
Arm/Group | SAP + Group Education | SAP + Standard Education | CSII + Group Education | CSII + Standard Education
Number analyzed (Participants) | 19 | 16 | 23 | 19
events per month | 0 (0) | 0 (0) | 0 (0) | 0 (0)

3. Secondary Outcome: Quality of Life (ADDQoL Questionnaire)
Description: Will be assessed QoL changes during the study and differences of these changes between groups.
  ADDQoL Questionnaire includes 2 general scales and 18 specific scales. 2 general scales represent the general QoL and diabetes - dependent QoL (scales varies from -3 (worse) to +3 (better)). 18 specific scales represent the impact of diabetes on certain QoL parameters: working life, family life, social life, sex life, physical appearance, do physically, leisure, travel, confidence in ability, motivation, society reaction, future, finances, dependence, living conditions, freedom to eat, other's , freedom to drink. All scales varies from -9 (worse) to +9 (better).
Time Frame: 4 month after CSII initiation
Population: Patients from structured education group completed the QoL Questionnaires prior to education and 4 months after transferring to CSII. Patients from the control group completed (standart education) the Questionnaires during the enrollment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | SAP + Group Education | SAP + Standard Education | CSII + Group Education | CSII + Standard Education
Number analyzed (Participants) | 19 | 16 | 23 | 19
units on a scale
  Working life (ADDQoL) | -1.68 (1.7) | -1.08 (2.19) | -1.09 (1.44) | -2.59 (2.39)
  Family life (ADDQoL) | -0.74 (3.07) | -1.08 (2.19) | -1.09 (1.44) | -2.59 (2.39)
  Social life (ADDQoL) | -0.37 (0.76) | -1.67 (2.35) | -0.09 (0.42) | -1.53 (2.8)
  Sex life (ADDQoL) | -0.89 (1.29) | -1.33 (1.92) | -0.27 (0.7) | -1.94 (2.11)
  Physical appearance (ADDQoL) | -1.0 (1.37) | -0.83 (1.27) | -0.61 (1.23) | -1.47 (2.06)
  Do physically (ADDQoL) | -2.47 (2.04) | -2.50 (2.28) | -1.35 (1.03) | -3.53 (2.93)
  Holidays/leisure (ADDQoL) | -1.32 (1.89) | -1.75 (2.86) | -0.7 (1.55) | -2.11 (2.69)
  Travel (ADDQoL) | -1.32 (1.53) | -1.67 (3.03) | -0.96 (1.58) | -2.32 (2.91)
  Confidence in ability (ADDQoL) | -1.32 (1.45) | 1.50 (1.73) | -0.65 (0.88) | -2.16 (2.34)
  Motivation (ADDQoL) | -0.53 (1.22) | -0.33 (3.47) | -0.13 (1.01) | -0.63 (3.42)
  Society reaction (ADDQoL) | 0 (0) | -0.50 (1.24) | -0.04 (0.47) | -0.79 (1.65)
  Future (ADDQoL) | -2.21 (2.3) | -4.42 (3.34) | -1.74 (2.26) | -4.11 (2.85)
  Finances (ADDQoL) | -1.05 (2.55) | -1.75 (1.71) | -1.30 (1.79) | -2.89 (2.92)
  Dependence (ADDQoL) | -0.42 (0.84) | -1.83 (2.48) | -0.36 (1.05) | -1.21 (2.07)
  Living conditions (ADDQoL) | -0.11 (1.2) | -0.25 (1.22) | -0.18 (0.59) | -0.74 (1.56)
  Freedom to eat (ADDQoL) | -0.95 (1.31) | -3.50 (3.53) | -1.86 (1.90) | -2.95 (2.34)
  Other's fuss (ADDQoL) | -0.47 (1.02) | -1.17 (1.99) | -0.50 (1.10) | -0.95 (2.55)
  Freedom to drink (ADDQoL) | -1.11 (1.63) | -1.58 (2.12) | -1.09 (1.38) | -1.89 (2.18)
  Present QoL (ADDQoL) | 1.00 (1.05) | 0.83 (1.34) | 1.09 (0.79) | 1.0 (1.0)
  Diabetes-related QoL (ADDQoL) | -1.32 (1.0) | -1.58 (1.0) | -1.13 (1.06) | -1.74 (0.87)

4. Secondary Outcome: Nonsevere Hypoglycaemia Frequency
Description: Nonsevere hypoglycemia is defined аs an episode of a blood glucose value of less than 70 mg per deciliter (3.9 mmol per liter). All hypoglycaemia episodes was reported in patients dairies and then will be assessed and compared between groups.
Time Frame: within 4 month of the study
Measure: Mean (Standard Deviation); unit: events per day
Arm/Group | SAP + Group Education | SAP + Standard Education | CSII + Group Education | CSII + Standard Education
Number analyzed (Participants) | 19 | 16 | 23 | 19
events per day | 0.13 (0.43) | 0.49 (0.91) | 0.43 (0.72) | 0.004 (0.06)

5. Secondary Outcome: Glycaemic Variability
Description: Several glucose variability scores was assessed: SD, MAGE, MODD, LI, HBGI, LBGI, MAG. For SAP users glucose variability scores were calculated from CGM data. For CSII users with SMBG only glucose variability scores were calculated from "bolus calculator" (Bolus Wizard) data.
Time Frame: within 4 month of the study
Reporting Status: Not Posted, anticipated posting 2015-11

6. Secondary Outcome: Treatment Compliance ( Frequency of SMBG and Bolus Calculator Use)
Description: Treatment compliance evaluation was based on frequency of SMBG and bolus calculator use as one of the factors mediating achievement of target plasma glucose level.
Time Frame: within 4 month of the study
Measure: Mean (Standard Deviation); unit: events
Arm/Group | SAP + Group Education | SAP + Standard Education | CSII + Group Education | CSII + Standard Education
Number analyzed (Participants) | 19 | 16 | 23 | 19
events
  frequency of SMBG | 6.7 (3.6) | 7.1 (6.2) | 4.6 (2.1) | 3.6 (2.4)
  frequency of bolus calculator use | 6.0 (2.7) | 5.4 (3.2) | 6.9 (3.2) | 4.8 (2.8)

7. Secondary Outcome: Quality of Life (SF36 Questionnaire)
Description: We assessed QoL changes during the study and differences of these changes between groups.
  SF-36 questionnaire enabling evaluation of patient's satisfaction with his health status and certain emotional characteristics. 36 items of the Questionnaire are grouped in 8 scales. Each scale ranges from 0 to 100, the latter representing full health.
Time Frame: 4 months after CSII initiation
Population: as for outcome 3
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | SAP + Group Education | SAP + Standard Education | CSII + Group Education | CSII + Standard Education
Number analyzed (Participants) | 19 | 16 | 23 | 19
units on a scale
  Physical Functioning | 95 [85 to 100] | 85 [70 to 95] | 95 [90 to 100] | 95 [85 to 100]
  Role-Physical Functioning | 88 [63 to 100] | 100 [38 to 100] | 100 [75 to 100] | 75 [75 to 100]
  Bodily Pain | 100 [84 to 100] | 63 [42 to 92] | 100 [84 to 100] | 84 [62 to 100]
  General Health | 67 [60 to 72] | 67 [15 to 87] | 67 [57 to 82] | 61 [37 to 67]
  Vitality | 70 [55 to 80] | 72.5 [33 to 80] | 65 [60 to 75] | 60 [40 to 75]
  Social Functioning | 88 [75 to 100] | 68.8 [50 to 88] | 88 [63 to 100] | 75 [63 to 88]
  Role Emotional | 100 [67 to 100] | 83 [67 to 100] | 100 [67 to 100] | 67 [33 to 100]
  Mental Health | 72 [62 to 80] | 72 [54 to 76] | 68 [60 to 84] | 60 [40 to 76]

ADVERSE EVENTS:
Arm/Group | SAP + Group Education | SAP + Standard Education | CSII + Group Education | CSII + Standard Education
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/16 | 0/23 | 0/19
Other Adverse Events (participants affected / at risk) | 0/19 | 0/16 | 0/23 | 0/19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes